CLINICAL TRIAL: NCT01420653
Title: Maxigesic 325 Acute Dental Pain Study: A Double-blind, Placebo-controlled, Randomized, Parallel Group Comparison of the Effects of Maxigesic 325 Versus Acetaminophen, Ibuprofen and Placebo in Participants With Acute Dental Pain
Brief Title: Maxigesic 325 Acute Dental Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFT-MX-6
Record Dates: First submitted 2011-08-16; First posted 2011-08-22 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2015-01

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Maxigesic 325 (Experimental): Acetaminophen 325mg + ibuprofen 97.5mg per tablet, two tablets every 6 hours, orally
  Interventions: Drug: Maxigesic 325
- Acetaminophen (Active Comparator): Acetaminophen 325mg per tablet (standard dose acetaminophen), two tablets every 6 hours, orally
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): Ibuprofen 97.5mg per tablet (i.e. low dose ibuprofen), two tablets every 6 hours, orally
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo tablets, every 6 hours, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maxigesic 325 — Maxigesic USA (acetaminophen 325 mg + ibuprofen 97.5mg), three tablets four times a day with food for 48 hours
  Other Names: Maxigesic
  Arms: Maxigesic 325
Drug: Acetaminophen — Acetaminophen 325 mg, 3 tablets four times a day, with food for 48 hours
  Other Names: paracetamol
  Arms: Acetaminophen
Drug: Ibuprofen — Ibuprofen 97.5mg, three tablets four times a day, with food for 48 hours.
  Arms: Ibuprofen
Drug: Placebo — placebo, three tablets four times a day, with food for 48 hours
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the analgesic effects of Maxigesic USA are greater than acetaminophen, ibuprofen or placebo.

DETAILED DESCRIPTION:
The combination of 500mg acetaminophen and 150mg ibuprofen has been shown to improve analgesia compared with the individual components, when given as 2 tablets (i.e. total of 1,000/300 mg) 4 times a day.

Recent concerns over the safety of acetaminophen have led to some regulatory agencies restricting the maximum dose of acetaminophen per tablet to 325 mg, while maintaining the maximum daily dose of 4000mg per day.

A dosing regimen of three tablets of Maxigesic 325 four times a day gives a total daily dose of 3900mg acetaminophen and 1170mg ibuprofen.

The primary objective of the study is to compare time-adjusted SPID of the VAS pain intensity scores up to 48 hours after the first dose of study medication among the four study groups.

Secondary objectives are:

To compare the time to onset of pain relief after the first dose of study drug defined as (i) perceptible and (ii) meaningful pain relief among the four study groups using the two stopwatch method.

To compare the maximum VAS pain scores up to 48 hours after the first dose of study medication among the four study groups.

To compare the response rates (response rate to be defined as the percentage of participants who reduce their pain intensity scores by at least 50% compared with the baseline VAS measure) among the four study groups.

To compare the time to peak reduction in VAS pain intensity scores following the first dose of study medication among the four study groups.

To compare the time to requirement for rescue medication among the four study groups.

To compare the percentage of participants who use rescue medication among the four study groups.

To compare the amount of rescue medication used (defined as number of tablets) among the four study groups.

To compare the categorical global pain rating among the four study groups.

Safety:

To compare adverse event rates for the 48-hour study period and up to Day 30 among the four treatment groups.

To compare the incidence of known specific NSAID and paracetamol side effects (e.g. GI ulceration or bleeding, indigestion/stomach pain, post-operative bleeding, bronchospasm, skin rashes, water retention, renal failure, thromboembolic events and evidence of clinical hepatitis) during the 48-hour study period and up to Day 30 among the four study groups.

Planned hospital admissions and/or surgical operations for an illness or disease which existed before the study drug was given or the participant was randomized in the study will not be considered adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent before initiation of any study-related procedures.
* Males and females aged at least 10 years and not more than 60 years old on the day of consent.
* Undergoing dental surgery for the extraction of at least 2 impacted third molar teeth.
* A resting VAS pain intensity score at baseline (within 6 hours after the completion of surgery) of greater than or equal to 40 mm on a 100 mm VAS scale with 0 = no pain and 100 = worst pain imaginable.

Exclusion Criteria:

* Has taken any NSAID or acetaminophen within 12 hours prior to the stat of surgery other than asprin less than or equal to 150 mg/day
* Subjects who have received any anaesthetics within 24 hours prior to surgery
* Hypersensitivity to opioids
* Known to be pregnant or possibly pregnant
* Women of childbearing potential who are unwilling to take adequate contraceptive precautions, i.e., hormonal contraceptive, an intrauterine device, double-barrier method, or abstinence. A women of childbearing potential is defined as any female who is less than 2 years post-menopausal or has not undergone a partial or total hysterectomy or surgical sterilization, e.g. bilateral tubal ligation, bilateral oophorectomy.
* Women of childbearing potential who are unwilling to undergo an urine pregnancy test.
* Suffering from a neurological disorder relating to pain perception or any acute or chronic condition that, in the opinion of the investigator, makes the subject unsuitable from an efficacy or safety perspective.
* In the opinion of the investigator, unable to understand the visual analogue pain score or comply with the protocol requirements.
* Currently, or in the last 30 days, has been in a clinical trial involving another study drug.
* Currently treated with an ACE inhibitor, warfarin, steroid (other than nasal steroids or topical steroids with the approval of the investigator) cyclosporin, tacrolimus or methotrexate, or any other medication felt by the investigator to interfere with safety or efficacy evaluations.
* Participant weight < 50 kg or > 120 kg.
* Has a history of drug or alcohol abuse.
* Suffering from any other disease or condition which, in the opinion of the investigator, means that it would not be in the participants best interests to participant in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Currie, Doctor, Principal Investigator — Clinical Trial New Zealand
Locations (4):
- Premier Research, Austin, Texas, United States
- New Zealand (3):
  - Clinical Trial New Zealand, Hamilton, Waikato Region
  - Clinical Solutions Ltd., Auckland
  - Southern Clinical Trials, Christchurch

REFERENCES:
- [Derived] Daniels SE, Atkinson HC, Stanescu I, Frampton C. Analgesic Efficacy of an Acetaminophen/Ibuprofen Fixed-dose Combination in Moderate to Severe Postoperative Dental Pain: A Randomized, Double-blind, Parallel-group, Placebo-controlled Trial. Clin Ther. 2018 Oct;40(10):1765-1776.e5. doi: 10.1016/j.clinthera.2018.08.019. Epub 2018 Sep 21. PMID 30245281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 455 Subjects have been consented and screened, out of which 47 subjects were screening failures and did not receive the first dose of study medication.
  Among 408 subjects, 273 subjects enrolled from New Zealand sites and 135 subjects enrolled from USA site from May 2013 to Jan 2015.
Period: Overall Study
Arm/Group | Maxigesic 325 | Acetaminophen | Ibuprofen | Placebo
Started | 110 | 111 | 112 | 75
Completed | 107 | 108 | 108 | 68
Not Completed | 3 | 3 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maxigesic 325 | Acetaminophen | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 110 | 111 | 112 | 75 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (7.0) | 25.0 (6.9) | 24.3 (5.9) | 24.3 (6.3) | 24.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 76 | 82 | 48 | 275
  Male | 41 | 35 | 30 | 27 | 133
Region of Enrollment [Number; unit: participants]
  New Zealand | 73 | 75 | 75 | 50 | 273
  United States | 37 | 36 | 37 | 25 | 135

OUTCOME MEASURES:

1. Primary Outcome: SPID (Summed Pain Intensity Differences)
Description: The time-adjusted Summed Pain Intensity Differences (SPIDs) of the VAS pain intensity scores up to 48 hours after the first dose of study medication.
  This was calculated from the visual analogue scale (VAS) pain intensity scores recorded during the 48 hours double blind treatment period, with the last measure taken just prior to the final dose of blinded study medication. The visual analogue scale is 100mm long with 0= no pain and 100=worst pain imaginable. The Visual Analogue Scale It is expected that treatments which can provide superior analgesic effect will demonstrate a greater Summed Pain Intensity Difference.
Time Frame: 48 hours afte the first dose
Population: Primary Efficacy Endpoint was analyzed in ITT population (subjects who have been randomized and received the first dose of study medication)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Maxigesic 325 | Acetaminophen | Ibuprofen | Placebo
Number analyzed (Participants) | 110 | 111 | 112 | 75
score on a scale | 31.56 (1.94) | 17.71 (1.89) | 23.18 (1.89) | 14.86 (2.26)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events were collected from the randomization to the follow up telephone contact made at 30 days after the surgery (Surgery Day is Day 1)
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information is the same as the one from the clinicatrials.gov.
Arm/Group | Maxigesic 325 | Acetaminophen | Ibuprofen | Placebo
All-Cause Mortality (participants affected / at risk) | 1/110 | 0/111 | 0/112 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/110 | 0/111 | 0/112 | 0/75
Other Adverse Events (participants affected / at risk) | 41/110 | 54/111 | 40/112 | 38/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maxigesic 325 (N=110) | Acetaminophen (N=111) | Ibuprofen (N=112) | Placebo (N=75)
Death due gun shot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The death was due to the gunshot wound (homicide) occurred during 30 days follow up period and not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maxigesic 325 (N=110) | Acetaminophen (N=111) | Ibuprofen (N=112) | Placebo (N=75)
Nausea (Gastrointestinal disorders) | 15 (18) | 19 (21) | 15 (15) | 17 (21)
Vomiting (Gastrointestinal disorders) | 9 (10) | 14 (17) | 5 (6) | 7 (8)
Headache (Nervous system disorders) | 8 (10) | 9 (10) | 9 (9) | 7 (8)
Facial swelling (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10) | 8 (8) | 5 (6)
Diziness (Nervous system disorders) | 4 (4) | 5 (5) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No